CLINICAL TRIAL: NCT05245097
Title: Mitigation of Major Hip Injury Due to Fall in an At-Risk, Older Adult Population With a Wearable Smart Belt
Brief Title: Mitigation of Major Hip Injury Due to Fall With a Smart Belt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ActiveProtective Technologies, Inc (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COP-0001
Record Dates: First submitted 2022-01-29; First posted 2022-02-17 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Hip Injuries; Fractures, Hip; Fall Injury; Fall Risk; Osteoporosis; Osteoporosis Risk
Keywords: Fall risk; Fall injury; Major hip injury; Hip fracture
MeSH Terms: conditions — Hip Injuries; Hip Fractures; Osteoporosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Intervention Group (Experimental): The intervention group will be assigned a Tango Belt to be worn around the waist for up to 24 hours a day (removed for bathing, charging of device and upon request) for 6 months. The Tango Belt (the "Device") is a wearable belt designed to enable safer mobility of geriatric individuals (≥ 65 years of age) at risk for fall injury by mitigating major hip injuries due to falls by deploying an airbag around the hips upon sensing a serious hip-impacting fall-in-progress to protect the hips from ground impact forces.
  Interventions: Device: Tango Belt; Other: Standard of Care (SOC)
- Control Group (Other): The clinical site's electronic medical record (EMR) database will be reviewed determine their long-term care patient population's initial eligibility for meeting the study inclusion criteria beginning at the time frame 6 months prior to the institutional review board (IRB) approval date. Subjects eligible for the control group must meet the requirements of the inclusion and exclusion criteria except for the waist circumference and need for consent. Eligible subjects' electronic health records will be mined for the baseline, midpoint, and final study metrics.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Device: Tango Belt — The Tango Belt is a patient-contacting electronic device made out of medical grade plastics and biocompatible fabrics worn around the waist. The Tango Belt contains a fall-in-progress detection algorithm which can detect a serious hip-impacting fall-in-progress using built-in sensors and deploy an automotive-grade cold-gas airbag to protect the hips from ground impact forces. When connected to Wi-Fi, the Tango Belt can send automated fall and impact alerts to caregivers and Healthcare Providers (HCPs) while recording motion and event data, which can then be analyzed for usage-based metrics viewable via a companion mobile app and/or desktop app. Alerts are sent in the form of short message service (SMS) texts and emails to alert recipients designated in the mobile or desktop Companion App. The Tango Belt can also detect non-serious hip-impacting or non-hip impacting falls in which the wearer may have incurred a minor injury (i.e., not a major hip injury) and/or may be unable to get up.
  Arms: Intervention Group
Other: Standard of Care (SOC) — The standard of care (SOC) in the US for managing the fall risk of geriatric patients is the CDC's Stopping Elderly Accidents, Deaths, and Injuries (STEADI) initiative, which implements the America and British Geriatric Societies'' Clinical Practice Guidelines for fall risk management. The STEADI algorithm consists of tools and resources for healthcare providers for fall risk screening, assessment, and interventioniv,v. Screening and assessment includes identifying fall history and modifiable factors related to fall and fall injury risk (e.g. fear of falling, gait, strength, balance, medications, comorbidities, etc.); then interventions to reduce the fall and fall injury risk are applied based upon assessment findings, and can include physical therapy, medication adjustments, patient education, bed and chair alarms, bed rails, etc.

SUMMARY:
Multi-center, comparative, non-significant risk adaptive study with retrospective controls.

After providing informed consent and being screened for eligibility, intervention subjects will be prescribed and provided an appropriately sized Tango Belt. The subject must demonstrate a minimum of 64% adherence to the use of the Tango Belt within 14 days of initiation to fully enroll in the study. Upon demonstration of at least minimum adherence, the subject will be provided the Tango Belt to wear continuously for at least 6 months, except during bathing, device charging, and as deemed by clinical staff.

The study will investigate the safety and effectiveness of the Tango Belt with the primary and secondary endpoints being taken every 3 months and at the end of the study run time from the electronic medical record. Additionally, ancillary endpoints on adverse events and device performance will be gathered.

DETAILED DESCRIPTION:
This is a multi-center, comparative, adaptive, non-significant risk clinical trial conducted in the United States to assess the safety and efficacy of the Tango Belt within senior care settings. Effectiveness of the Tango Belt will be determined by analysis of evidence for the Tango Belt as an adjunctive intervention to the standard-of-care (SOC) to mitigate major hip injuries from falls in an older adult population at-risk for fall injury as the primary endpoint. Performance of the Tango Belt to mitigate fall injuries that result in hip fracture, emergency room visits, and hospitalizations will be secondary endpoints. The performance of the device is determined by the comparison of the proportion of fall-related major hip injuries in the intervention group as compared to the proportion of fall-related major hip injuries in a retrospective control group utilizing only SOC. SOC utilization will be verified for each clinical site enrolled. An adaptive trial design will be utilized to allow an initial efficacy target to be evaluated at 6 months; if the initial target is not met, then a second cohort of sites and subjects will be enrolled for an additional 6 months to allow a lower efficacy target to be evaluated.

Safety of the device will be determined by analysis of adverse events as an ancillary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older;
2. Have experienced a fall-related fracture after age 50 -OR- Have experienced one or more falls in the 12-months prior to consent and have a diagnosis of osteoporosis, osteopenia, or prescribed osteoporosis medication.
3. Independently or with staff or caregiver assistance, able to transfer between surfaces (e.g., to or from a bed, chair, wheelchair, toilet, standing position) or walk or move between locations (use of an assistive device such as a walker is acceptable);
4. Have a waist circumference between 29 - 50 inches (63.5 - 127 cm);
5. Able to comply with required study procedures and follow-up schedule as determined by the Study Investigator;
6. Are under the care of the Investigational organization;
7. Provides consent or their legally authorized representative provides consent on subject's behalf

Exclusion Criteria:

1. Age 64 years or less;
2. Participation in a different clinical investigation that can conflict with this clinical study as determined by the Study Investigator and approved by the Sponsor;
3. Total dependence on staff or caregiver assistance to be able to transfer between surfaces (e.g., to or from a bed, chair, wheelchair, toilet, standing position) and walk and move between locations;
4. Use of other devices or interventions outside of SOC (Standard of care) for fall risk management during study participation without Sponsor approval;
5. Unable to comply with required study procedures and follow-up schedule as determined by the Study Investigator;
6. Does not provide consent, or legally authorized representative does not provide consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 471 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Stefanacci, DO, MGH,MBA, AGSF, CMD, Principal Investigator — ActiveProtective Technologies, Inc
Locations (10):
- United States (10):
  - Revere Court of Sacramento, Sacramento, California
  - Holy Redeemer Health System, Bensalem, Pennsylvania
  - Foulkeways at Gwynedd, Gwynedd, Pennsylvania
  - Country Meadows Hershey, Hershey, Pennsylvania
  - Meadowood Senior Living, Lansdale, Pennsylvania
  - Camilla Hall, Malvern, Pennsylvania
  - Chandler Hall Health Services, Newtown, Pennsylvania
  - The Heritage of Green Hills, Shillington, Pennsylvania
  - Country Meadows Wyomissing, Wyomissing, Pennsylvania
  - Country Meadows of York-South, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CDC Facts About Falls. (2021, August 6). Centers for Disease Control and Prevention. https://www.cdc.gov/falls/facts.html
- [Background] Bergen G, Stevens MR, Burns ER. Falls and Fall Injuries Among Adults Aged >/=65 Years - United States, 2014. MMWR Morb Mortal Wkly Rep. 2016 Sep 23;65(37):993-998. doi: 10.15585/mmwr.mm6537a2. PMID 27656914
- [Background] Florence CS, Bergen G, Atherly A, Burns E, Stevens J, Drake C. Medical Costs of Fatal and Nonfatal Falls in Older Adults. J Am Geriatr Soc. 2018 Apr;66(4):693-698. doi: 10.1111/jgs.15304. Epub 2018 Mar 7. PMID 29512120
- [Background] Panel on Prevention of Falls in Older Persons, American Geriatrics Society and British Geriatrics Society. Summary of the Updated American Geriatrics Society/British Geriatrics Society clinical practice guideline for prevention of falls in older persons. J Am Geriatr Soc. 2011 Jan;59(1):148-57. doi: 10.1111/j.1532-5415.2010.03234.x. PMID 21226685
- [Background] CDC STEADI - Older Adult Fall Prevention, Resource Algorithm for Fall Risk Screening, Assessment, and Intervention. 2019. Centers for Disease Control and Prevention. www.cdc.gov/steadi.
- [Background] Stefanacci RG, Haimowitz D. Stand by me--preventing falls. Geriatr Nurs. 2012 Mar-Apr;33(2):134-6. doi: 10.1016/j.gerinurse.2012.02.003. No abstract available. PMID 22464055
- [Background] Kannus P, Parkkari J, Niemi S, Pasanen M, Palvanen M, Jarvinen M, Vuori I. Prevention of hip fracture in elderly people with use of a hip protector. N Engl J Med. 2000 Nov 23;343(21):1506-13. doi: 10.1056/NEJM200011233432101. PMID 11087879
- [Background] Parker MJ, Gillespie WJ, Gillespie LD. Effectiveness of hip protectors for preventing hip fractures in elderly people: systematic review. BMJ. 2006 Mar 11;332(7541):571-4. doi: 10.1136/bmj.38753.375324.7C. Epub 2006 Mar 2. PMID 16513687
- [Background] Bulat T, Powell-Cope G, Rubenstein L. Perceived Barriers and Facilitators for the Use of External Hip Protectors. Gerontological Journal. June 2004, Vol 3, No1.
- [Background] Parkkari J, Heikkila J, Kannus IP. Acceptability and compliance with wearing energy-shunting hip protectors: a 6-month prospective follow-up in a Finnish nursing home. Age Ageing. 1998 Mar;27(2):225-9. doi: 10.1093/ageing/27.2.225. PMID 16296684
- [Background] Moreland B, Kakara R, Henry A. Trends in Nonfatal Falls and Fall-Related Injuries Among Adults Aged >/=65 Years - United States, 2012-2018. MMWR Morb Mortal Wkly Rep. 2020 Jul 10;69(27):875-881. doi: 10.15585/mmwr.mm6927a5. PMID 32644982
- [Background] Bhasin S, Gill TM, Reuben DB, Latham NK, Ganz DA, Greene EJ, Dziura J, Basaria S, Gurwitz JH, Dykes PC, McMahon S, Storer TW, Gazarian P, Miller ME, Travison TG, Esserman D, Carnie MB, Goehring L, Fagan M, Greenspan SL, Alexander N, Wiggins J, Ko F, Siu AL, Volpi E, Wu AW, Rich J, Waring SC, Wallace RB, Casteel C, Resnick NM, Magaziner J, Charpentier P, Lu C, Araujo K, Rajeevan H, Meng C, Allore H, Brawley BF, Eder R, McGloin JM, Skokos EA, Duncan PW, Baker D, Boult C, Correa-de-Araujo R, Peduzzi P; STRIDE Trial Investigators. A Randomized Trial of a Multifactorial Strategy to Prevent Serious Fall Injuries. N Engl J Med. 2020 Jul 9;383(2):129-140. doi: 10.1056/NEJMoa2002183. PMID 32640131
- [Background] Gill TM, Bhasin S, Reuben DB, Latham NK, Araujo K, Ganz DA, Boult C, Wu AW, Magaziner J, Alexander N, Wallace RB, Miller ME, Travison TG, Greenspan SL, Gurwitz JH, Rich J, Volpi E, Waring SC, Manini TM, Min LC, Teresi J, Dykes PC, McMahon S, McGloin JM, Skokos EA, Charpentier P, Basaria S, Duncan PW, Storer TW, Gazarian P, Allore HG, Dziura J, Esserman D, Carnie MB, Hanson C, Ko F, Resnick NM, Wiggins J, Lu C, Meng C, Goehring L, Fagan M, Correa-de-Araujo R, Casteel C, Peduzzi P, Greene EJ. Effect of a Multifactorial Fall Injury Prevention Intervention on Patient Well-Being: The STRIDE Study. J Am Geriatr Soc. 2021 Jan;69(1):173-179. doi: 10.1111/jgs.16854. Epub 2020 Oct 9. PMID 33037632
- [Background] Yang Y, Komisar V, Shishov N, Lo B, Korall AM, Feldman F, Robinovitch SN. The Effect of Fall Biomechanics on Risk for Hip Fracture in Older Adults: A Cohort Study of Video-Captured Falls in Long-Term Care. J Bone Miner Res. 2020 Oct;35(10):1914-1922. doi: 10.1002/jbmr.4048. Epub 2020 Jul 6. PMID 32402136
- [Background] Quigley P, Singhatat W, Tarbert R. Technology Innovation to Protect Hips from Fall-Related Fracture. 2019, Phys Med Rehabil Res. Vol 4. 104. DOI: 10.15761/PMRR.1000205
- [Background] Tarbert R, Singhatat W. Skilled Nursing Resident Adherence with Wearable Technology to Offer Safer Mobility and Decreased Fall Injuries. 2020. Journal of Pat Safety and Risk Man. DOI: 10.1177/2516043520979193
- [Derived] Stefanacci RG, Kinosian B. Mitigating Hip Injuries in High-Risk Older Adults: Clinical Evidence Supporting FDA Approval of a Novel Wearable Airbag Belt. J Am Med Dir Assoc. 2025 Nov;26(11):105851. doi: 10.1016/j.jamda.2025.105851. Epub 2025 Sep 10. PMID 40887039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The intervention group was recruited via clinical site health record review for the inclusion/exclusion criteria available and waist circumference obtained by sub-investigator on-site and offered informed consent. The control group was determined via historical clinical site health record review determining subject eligibility based on inclusion/exclusion criteria except waist circumference and did not need consent.
Pre-assignment Details: Intervention subjects initially enrolled (207) attempted a 14-day run-in period during which adherence to use of the study device was measured. 73 subjects who do not meet the run-in period requirement (64% adherence to wear) were withdrawn from the study resulting in 134 fully enrolled intervention group subjects.
Groups:
- Intervention Group: 134 patients were fully enrolled into the intervention group after achieving the minimum run-in adherence with the withdrawal of 73 patients prior to achieving or failing Run-In.
- Control Group: 264 retrospective control subjects were matched to the fully enrolled intervention group of 134.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 134 | 264
Completed | 79 | 246
Not Completed | 55 | 18
Not completed — Adverse Event | 13 | 2
Not completed — Protocol Violation | 8 | 6
Not completed — Withdrawal by Subject | 18 | 0
Not completed — Death | 6 | 7
Not completed — Physician Decision | 6 | 0
Not completed — Relocation | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: The intervention group subjects meeting the requirements of the inclusion and exclusion criteria and who consented to study enrollment, received Standard of Care (SOC) for managing fall risk as per the CDC's Stopping Elderly Accidents, Deaths, and Injuries (STEADI) initiative and were assigned a Tango Belt to be worn around the waist for up to 24 hours a day (removed for bathing, charging of device and upon request) for 6 months.
- Control Group: Control group subjects meeting the requirements of the inclusion and exclusion criteria (except for the waist circumference and need for consent) were identified via clinical site health records and received the standard of care (SOC) for managing fall risk as per the CDC's Stopping Elderly Accidents, Deaths, and Injuries (STEADI) initiative. Their falls and fall injuries were recorded for the 6 months following their retrospective enrollment date.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 134 | 264 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 87.3 (7.15) | 87.5 (6.40) | 87.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 209 | 311
  Male | 32 | 55 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 0 | 0 | 0
  Race: Asian | 1 | 4 | 5
  Race: Black or African American | 1 | 1 | 2
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 129 | 257 | 386
  Race: Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 134 | 264 | 398
Highest Mobility Level [Count of Participants; unit: Participants]
  Independent | 75 | 149 | 224
  Supervision | 24 | 44 | 68
  Limited Assist | 34 | 70 | 104
  Extensive Assist | 1 | 1 | 2
  Total Dependence | 0 | 0 | 0
Fall Risk Factor [Count of Participants; unit: Participants] | 125 | 249 | 374

OUTCOME MEASURES:

1. Primary Outcome: Major Hip Injuries Due to Serious Hip-impacting Fall
Description: The percent of subjects in the ITT population with major hip injuries due to serious hip-impacting falls.
Time Frame: 6 months
Population: The analysis population consists of all intervention population subjects who demonstrated at least 64% adherence to use of device during run-in period and the propensity matched historical controls.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Intervention Group: The intervention group was assigned a Tango Belt to be worn around the waist for up to 24 hours a day (removed for bathing, charging of device and upon request) for 6 months and received Standard of Care (SOC) for managing the fall risk of geriatric patients is the CDC's Stopping Elderly Accidents, Deaths, and Injuries (STEADI) initiative, which implements the America and British Geriatric Societies'' Clinical Practice Guidelines for fall risk management.
- Control Group: The control group received Standard of Care (SOC) for managing the fall risk of geriatric patients is the CDC's Stopping Elderly Accidents, Deaths, and Injuries (STEADI) initiative, which implements the America and British Geriatric Societies'' Clinical Practice Guidelines for fall risk management. Data points on falls and fall injuries were gathered via review of subject health records for their 6 month in-study time.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 134 | 264
percentage of participants | 1.1 [0.00 to 3.39] | 12.1 [8.44 to 16.68]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other — For the multiple imputation, a total of 50 imputed datasets will be calculated (Graham et al.). Fully conditional specification (FCS) discriminant function method will be used to impute missing primary endpoint using the baseline covariates of age, sex, race, ethnicity, mobility level, and BIMS Score. The FCS logistic method was replaced with the FCS discriminant function method due to a quasi-separation caused by only one observed primary endpoint event in the treatment group; p = 0.004, Regression, Logistic — The null hypothesis was tested at a one-sided 0.025 level of significance using a logistic regression analysis to compare treatment groups while controlling for propensity score

2. Secondary Outcome: Number of Hip Fractures Related to Fall
Description: The number of subjects in the ITT group with hip fractures related to a fall event.
Time Frame: 6 months
Population: The analysis population consisted of all intervention population subjects who demonstrate at least 64% adherence to use of device during run-in period (defined as wearing device for at least 1 hour per day for at least 9 of 14 days) and the propensity matched historical controls.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 134 | 264
participants | 3 [1 to 9] | 30 [21 to 42]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p = 0.003, Regression, Logistic — The hip fracture due to fall rate was compared between treatment groups using firth logistic regression while controlling for propensity score. A one-sided 0.025 level of significance was used
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.003, Regression, Logistic

3. Secondary Outcome: Number of Emergency Department Visits Related to Fall
Description: The number of subjects in the ITT group with emergency department visits related to fall.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 134 | 264
participants | 8 [3 to 15] | 47 [36 to 60]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.001, Regression, Logistic — The emergency department visit due to fall rate was compared between treatment groups using firth logistic regression while controlling for propensity score. A one-sided 0.025 level of significance was used; Subjects with multiple ED visits due to falls are only counted once

4. Secondary Outcome: Number of Hospitalizations Due to Fall
Description: The number of subjects in the ITT group admitted to a hospital due to fall.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 134 | 264
participants | 11 [6 to 19] | 50 [38 to 64]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority; p = 0.003, Regression, Logistic — The hospitalization due to fall rate was compared between treatment groups using firth logistic regression while controlling for propensity score. A one-sided 0.025 level of significance was used; Subjects with multiple hospitalizations due to falls are only counted once

5. Other Pre Specified Outcome: Number and Severity of Adverse Events
Description: An Adverse Event is any untoward medical occurrences in a patient or subject receiving an investigational medical device and does not necessarily have to have a causal relationship with the device under investigation. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical device whether or not considered related to the medical device. Any fall event is considered an AE for this study. A Severe Adverse Event is any AE that results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/ incapacity.
Time Frame: 6 months
Population: The safety population includes all subjects who were assigned a Tango Belt and attempted the run-in period.
Measure: Number; unit: Number of events
Groups:
- Safety Population: The Safety Population includes all intervention subjects that were offered the study device and entered into the run-in period (207) prior to full study enrollment after passing the adherence metric (134). This group was assigned a Tango Belt to be worn around the waist for up to 24 hours a day (removed for bathing, charging of device and upon request) for 6 months and received Standard of Care (SOC) for managing the fall risk of geriatric patients is the CDC's Stopping Elderly Accidents, Deaths, and Injuries (STEADI) initiative, which implements the America and British Geriatric Societies'' Clinical Practice Guidelines for fall risk management.
Arm/Group | Safety Population | Control Group
Number analyzed (Participants) | 207 | 264
Number of events
  Mild Severity Adverse event | 163 | 232
  Moderate Severity Adverse Event | 29 | 70
  Severe Severity Adverse Event | 27 | 66

6. Other Pre Specified Outcome: Number of Major Injuries Due to Fall
Description: The number of major injuries that were due to a fall.
Time Frame: 6 months
Measure: Number; unit: Major injuries due to fall
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 134 | 264
Major injuries due to fall | 7 | 67

7. Other Pre Specified Outcome: Rate of Fall Occurence
Description: The fall rate for the intervention and the control group
Time Frame: 6 months
Population: The fall rate ratio was compared between treatment groups using a Poisson regression model. Treatment was the independent variable and the log of total 180-day durations was the offset variable. The p-value corresponds to the beta coefficient on the treatment variable. A two-sided 0.05 level of significance was used.
Measure: Number; unit: Falls per 180-day duration
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 134 | 264
Falls per 180-day duration | 1.56 | 1.31

8. Other Pre Specified Outcome: Device Wear Adherence
Description: Adherence to wearing of the study device in days/month
Time Frame: 90 days and 180 days
Population: The study device was not offered to the control group and so device adherence was only measured for the intervention group.
Measure: Mean (Standard Deviation); unit: Tango Belt wear in Days/month
Arm/Group | Intervention Group
Number analyzed (Participants) | 134
Tango Belt wear in Days/month
  90 day: number analyzed (Participants) | 97
  90 day | 21.9 (6.08)
  180 day: number analyzed (Participants) | 79
  180 day | 20.1 (6.71)

9. Other Pre Specified Outcome: Device Wear Compliance
Description: Compliance to wearing of the study device in hours/day average
Time Frame: 6 months
Measure: Number; unit: hours/day in-study time
Arm/Group | Intervention Group
Number analyzed (Participants) | 134
hours/day in-study time | 5.9

10. Other Pre Specified Outcome: Accuracy of Device Fall Discrimination
Description: Rate of airbag deployments that occurred while an intervention subject was not experiencing a serious hip-impacting fall.
Time Frame: 6 months
Measure: Number; unit: false positives per 1000 person-days
Arm/Group | Safety Population
Number analyzed (Participants) | 207
false positives per 1000 person-days | 1.59

11. Other Pre Specified Outcome: Accuracy of Study Device Airbag Deployment
Description: Accuracy of the study device airbag deployment as designed is demonstrated in the number of hip fractures that occurred by intervention subjects wearing the device during serious hip-impacting falls.
Time Frame: 6 months
Population: The adherence population includes all subjects in the PP population excluding those subjects who were not actually wearing Tango Belt when the primary effectiveness endpoint was experienced.
Measure: Count of Participants; unit: Participants
Groups:
- The Adherence Population: The adherence population includes all subjects in the ITT who additionally met all study eligibility criteria, have available study data for the study endpoint and do not have a major protocol violation that effects primary effectiveness and the propensity matched historical controls. This population also excludes those subjects who were not actually wearing Tango Belt when the primary effectiveness endpoint was experienced.
Arm/Group | The Adherence Population
Number analyzed (Participants) | 132
Participants | 0

12. Other Pre Specified Outcome: Balance Confidence Score Changes
Description: Short version of the Falls Efficacy Scale International (where applicable for those deemed able to take the questionnaire (BIMS of 13-15)) to offer level of balance confidence as defined by the scale (range from 7 (no concern about falling) to 28 (severe concern about falling).
Time Frame: 6 months
Population: The number of intervention subjects changed as the study time line proceeded and some intervention subjects exited prior to the 90 day and 180 day.
Measure: Mean (Standard Deviation); unit: FES-I Short Version Score
Arm/Group | Intervention Group
Number analyzed (Participants) | 134
FES-I Short Version Score
  Baseline: number analyzed (Participants) | 63
  Baseline | 15.3 (4.29)
  90 day: number analyzed (Participants) | 48
  90 day | 15.4 (4.16)
  180 day: number analyzed (Participants) | 44
  180 day | 14.7 (4.68)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for all study subjects within their respective 6 month in-study timeframe.
Description: An Adverse Event (AE) is any untoward medical occurrences in a patient or subject receiving an investigational medical device and does not necessarily have to have a causal relationship with the device under investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medical device whether or not considered related to the medical device. Any fall event is considered an AE for this study. Severity assessed by investigator.
Arm/Group | Safety Population | Control Group
All-Cause Mortality (participants affected / at risk) | 6/207 | 7/264
Serious Adverse Events (participants affected / at risk) | 33/207 | 66/264
Other Adverse Events (participants affected / at risk) | 67/207 | 152/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=207) | Control Group (N=264)
Fall with Fracture (Musculoskeletal and connective tissue disorders) | 6 (6) | 57 (59) — A fall occurred with a related fracture outcome
Infection (Infections and infestations) | 4 (4) | 1 (1)
Dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other (General disorders) | 23 (23) | 7 (7) — Chronic vascular, cardiologic, pulmonary disease exacerbations and infections
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=207) | Control Group (N=264)
Fall Event (Musculoskeletal and connective tissue disorders) | 44 (145) | 119 (276) — Multiple subjects suffered multiple falls during their in-study phase which created a number of events higher than the number of group members.
Discomfort (Skin and subcutaneous tissue disorders) | 25 (25) | 40 (51)
Soreness (Musculoskeletal and connective tissue disorders) | 4 (4) | 13 (13)
abrassion (Skin and subcutaneous tissue disorders) | 9 (10) | 25 (25)
confusion (Psychiatric disorders) | 6 (7) | 14 (18)
Laceration (Skin and subcutaneous tissue disorders) | 14 (15) | 32 (36)
Other (General disorders) | 24 (39) | 25 (29) — Chronic pulmonary, venous and cardiac syndrome exacerbations or infections

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05245097/Prot_SAP_ICF_001.pdf